CLINICAL TRIAL: NCT02993796
Title: The Institute for Myelin and Glia Exploration's Clinical Database of Patients With Krabbe Disease, A World-Wide Registry
Brief Title: Krabbe Disease Global Patient Registry
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); Lysosomal Disease Network (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thomas J. Langan, Principal Investigator, State University of New York at Buffalo
Other Study IDs: RDCRN6726; 1R01HD104814-01A1 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-15 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Krabbe Disease
Keywords: Krabbe disease; globoid cell leukodystrophy; galactosylceramide lipidosis; sphingolipidosis
MeSH Terms: conditions — Leukodystrophy, Globoid Cell; Sphingolipidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a clinical database of individuals diagnosed with Krabbe disease in order to determine which symptoms herald the onset of clinical disease in the various phenotypes of Krabbe disease; to determine whether level of GALC enzyme activity, or a specific genetic mutation predict the clinical course; and to determine which neurodiagnostic tests predict onset and/or severity of the disease.

DETAILED DESCRIPTION:
The purported incidence of Krabbe disease is 1/250,000 live births. It is believed that 80-90% of affected children will have the early-infantile form of the disease. Other forms of the disease, however, occur throughout life. Unfortunately neither enzyme activity levels nor specific genetic mutation reliably predict phenotype. Since the only treatment for Krabbe disease is bone marrow transplantation, it is crucial to be able to identify prognostic factors, which will accurately predict the disease course. At this time the medical literature is limited regarding the clinical signs and symptoms of the later-onset forms of Krabbe disease, as well as their age of onset, and survival of these individuals.

Early-infantile Krabbe disease has a uniformly fatal outcome if untreated, and later-onset forms remain at-risk for developing symptoms. The only available treatment, pooled cord-blood transplantation, has a 10-20% mortality rate.

The vast majority of children who screen positively for Krabbe disease during newborn screening have an uncertain prognosis. No single diagnostic test available currently can accurately predict the onset of symptoms. Consequently, improved phenotypic understanding will enhance the diagnostic paradigm for Krabbe disease, and will facilitate more timely diagnosis and treatment.

The information collected in the registry will be used to improve accuracy of diagnosis, and to prevent children who are not destined to develop Krabbe from being subjected unnecessarily to treatment.

The hypotheses to be tested include:

* a detailed database will broaden phenotypic understanding of Krabbe disease;
* new therapies will result from better phenotypic understanding of this disorder.

A questionnaire will be collected at time of enrollment with information pertaining to an individual affected by Krabbe disease. Clinical information to be collected will include: age at onset of symptoms; type of symptoms; age at diagnosis; level of GALC enzyme activity; identification of the specific genetic mutation; results of any available brain MRI imaging evaluations; results of any available spinal fluid protein analyses; results of any available brainstem auditory evoked response evaluations; results of any available visual evoked response evaluations; and results of any available nerve-conduction-velocity studies. If possible, CD-ROMs containing the imaging data and physician reports of brain MRI imaging evaluations will be obtained. Potential prognostic indicators based on molecular genetic results, GALC enzyme level, detected potential biomarkers, and neurodiagnostic testing will be analyzed. Information on the status of participant's general health, disease progression, impact of the disease, neurologic symptoms, and developmental milestones will be collected through follow-up phone calls with parents or caregivers.

After de-identification, the data will be entered into the Krabbe clinical database at the University at Buffalo's Center of Excellence in Bioinformatics, and/or the Population Health Observatory on the South Campus, and/or the Longitudinal Pediatric Data Resource, a tool provided by the Newborn Screening Translational Research Network.

ELIGIBILITY:
Inclusion Criteria:

* Anyone diagnosed with Krabbe disease
* Anyone at-risk for Krabbe disease
* Family members of someone diagnosed with, or at-risk for, Krabbe disease.

Exclusion Criteria:

* Anyone who is not diagnosed with, or at-risk for, Krabbe disease
* Anyone who is not a family member of someone diagnosed with, or at-risk for, Krabbe disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study seeks enrollment by anyone of any age or gender who has been diagnosed with Krabbe disease, and also:
  * Anyone at-risk for Krabbe disease
  * Family members of someone diagnosed with, or at-risk for, Krabbe disease. This may consist of adults unable to consent; individuals who are not yet adults; and pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | up to 5 years
  The longevity of participants will be recorded using their date of death, or conclusion of this study, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Langan, MD, Principal Investigator — Clinical Director, Clinical Research, Institute for Myelin and Glial Exploration
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data is input to the NIH-funded Rare Diseases Clinical Research Network's Data Management & Coordinating Center ("DMCC"). Eventually this data will become part of the database of Genotypes and Phenotypes ("dbGaP"), which is part of the National Center for Biotechnology Information, U.S. National Library of Medicine.

REFERENCES:
- [Background] Carter RL, Wrabetz L, Jalal K, Orsini JJ, Barczykowski AL, Matern D, Langan TJ. Can psychosine and galactocerebrosidase activity predict early-infantile Krabbe's disease presymptomatically? J Neurosci Res. 2016 Nov;94(11):1084-93. doi: 10.1002/jnr.23793. PMID 27638594
- [Background] Langan TJ, Barcykowski AL, Dare J, Pannullo EC, Muscarella L, Carter RL. Evidence for improved survival in postsymptomatic stem cell-transplanted patients with Krabbe's disease. J Neurosci Res. 2016 Nov;94(11):1189-94. doi: 10.1002/jnr.23787. PMID 27638603
- See also: Hunter James Kelly Research Institute, University at Buffalo - home page — http://hjkri.buffalo.edu/
- See also: Hunter's Hope Foundation, one of the funders of this research study - their home page — http://huntershope.org/
- See also: Newborn Screening Translational Research Network - their home page — https://www.nbstrn.org/
- See also: Eunice Kennedy Shriver National Institute of Child Health and Human Development — https://www.nichd.nih.gov/Pages/index.aspx
- See also: Rare Diseases Clinical Research Network, the funder of the Lysosomal Disease Network — https://www.rarediseasesnetwork.org/